CLINICAL TRIAL: NCT02327988
Title: Cryotherapy and Laser Therapy do Not Interfere in the Response to Eccentric Exercise-induced Muscle Damage: a Randomized Clinical Trial.
Brief Title: Cryotherapy and Laser Therapy on Muscle Damage
Acronym: CLMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Jamilson Simões Brasileiro, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 387.826
Record Dates: First submitted 2014-12-11; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Myalgia [C05.651.542]
Keywords: cryotherapy; laser therapy; eccentric exercise; delayed onset muscle soreness; muscle damage; dynamometry; electromyography
MeSH Terms: interventions — Cryotherapy; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cryotherapy (Experimental): To the cryotherapy group a 1kg ice pack was strapped over the entire brachial biceps muscle and adjacent muscles of the arm under study using a bandage, and the application lasted 25 minute laser
  Interventions: Other: Cryotherapy
- Laser therapy (Experimental): The laser therapy group received laser application to the muscle belly of the non-dominant upper limb brachial biceps at four different points.
  Interventions: Device: Laser therapy
- Control (No Intervention): The control group did not undergo any intervention and remained at rest for 25 minutes.

INTERVENTIONS:
Other: Cryotherapy
  Arms: Cryotherapy
Device: Laser therapy
  Arms: Laser therapy

SUMMARY:
This study propose investigate the effect of cryotherapy and laser therapy in response to strenuous exercise-induced muscle damage on the biceps brachii muscle (muscle of the arms). All the individuals underwent to an strenuous exercise protocol (2 series of 10 contractions of non-dominant elbow flexors) and three assessments (pre, post and 48hr after the exercise), composed of pain sensation, measure of the strength and muscle activation.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Aged between 18 and 28 years
* Healthy, considered active according to the International Physical Activity Questionnaire -Short Form (IPAQ)
* Engaging in physical activity involving upper limbs at least 2 times a week
* Exhibiting shoulder joint, elbow and non-dominant hand integrity
* Not having a history of osteo-myoarticular injuries in the assessed limb in the last 6 months, or neurological, visual and/or non-corrected auditory impairments.
* Furthermore they could not be allergic to ice (verified by the ice cube test) or any absolute contraindication for the use of laser (cancer and pregnancy).

Exclusion Criteria:

* Not understanding the commands given in the protocols and/or inadequate performance during assessments.

Ages: 18 Years to 28 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain sensation | Within the first 3 days
  Through the VAS (visual analogue scale).

SECONDARY OUTCOMES:
Strength | Within the first 3 days
  The strength will be measure through isokinetic dynamometry and the variables analyzed will be peak torque normalized for body weight and power.
Muscle activation | Within the first 3 days
  Measured by surface electromyography.